CLINICAL TRIAL: NCT02622724
Title: A Phase III Double-blind, Randomised, Parallel-Group Comparison of the Efficacy and Safety of FP-1201-lyo (Recombinant Human IFN Beta-1a) and Placebo in the Treatment of Patients With Moderate or Severe Acute Respiratory Distress Syndrome
Brief Title: Efficacy and Safety of FP-1201-lyo (Interferon Beta-1a) in Patients Having Acute Respiratory Distress Syndrome (ARDS)
Acronym: INTEREST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Day 90 results indicate IMP did not reduce mortality or ventilator free days
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FPCLI002; 2014-005260-15 (EudraCT Number)
Record Dates: First submitted 2015-11-24; First posted 2015-12-04 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: ARDS, human; Acute Respiratory Distress Syndrome; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FP-1201-lyo 10 μg (Experimental): FP-1201-lyo 10 μg (Interferon beta-1a) will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational product is lyophilisate for solution for injection which will be reconstituted in water for injection.
  Interventions: Drug: Interferon beta-1a
- FP-1201-lyo Placebo (Placebo Comparator): FP-1201-lyo Placebo will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational placebo product is lyophilisate for solution for injection which will be reconstituted in water for injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon beta-1a — Investigational drug
  Other Names: FP-1201-lyo; Traumakine; ATC code L03AB07
  Arms: FP-1201-lyo 10 μg
Drug: Placebo — Placebo for investigational drug
  Other Names: FP-1201-lyo Placebo
  Arms: FP-1201-lyo Placebo

SUMMARY:
In this study effectiveness and safety of a new drug FP-1201-lyo (recombinant human interferon beta-1a) is compared to placebo. Investigation is conducted with patients who have acute respiratory distress syndrome (ARDS). The new drug is expected to reduce the time which a patient need to be on the ventilator and improve patient's chances of survival. Currently there are no approved drugs for treating moderate or severe ARDS patients.

DETAILED DESCRIPTION:
This is a Phase III clinical study to investigate the efficacy and safety of FP-1201-lyo (recombinant human interferon [IFN] beta-1a) compared to placebo in patients diagnosed with moderate or severe acute respiratory distress syndrome (ARDS). Primary objective is to demonstrate the efficacy of FP-1201-lyo in improving the clinical course and outcome based on survival and need for mechanical ventilation. Currently there are no approved drugs for treating moderate or severe ARDS patients.

FP-1201-lyo is a lyophilised powder form of recombinant human IFN beta-1a reconstituted in water for injection and is administered intravenously.

Recombinant human IFN beta-1a is an approved treatment for patients for other indication and its safety profile in such patients is well characterised.

ELIGIBILITY:
Inclusion Criteria:

All patients must be intubated and mechanically ventilated to diagnose ARDS and be eligible for the study

1. Patient has a diagnosis of moderate or severe ARDS according to the Berlin definition of ARDS:

   * Acute onset of respiratory failure within 1 week of a known clinical insult or new or worsening respiratory symptoms
   * Respiratory failure associated with known ARDS risk factors and not fully explained by either cardiac failure or fluid overload (an objective assessment of cardiac failure or fluid overload is needed if no risk factors for ARDS [moderate or severe ARDS] are present)
   * Radiological abnormalities on chest X-ray or on computerised tomography scan, i.e., bilateral opacities that are not fully explained by effusions, nodules, masses or lobar/lung collapse
   * Hypoxaemia:

     * Moderate ARDS: PaO2/FiO2 >100 mmHg (>13.3 kPa) to ≤200 mmHg (≤26.6 kPa) with positive end expiratory pressure (PEEP) ≥5 cmH2O
     * Severe ARDS: PaO2/FiO2 ≤100 mmHg (≤13.3 kPa) with positive end expiratory pressure [PEEP] ≥5 centimeter of water [cmH2O]
2. The radiological and hypoxaemia criteria (1.3 and 1.4) must be met within the same 24-hour period. The time of onset of ARDS is when the last of the two specified ARDS criteria is met
3. Administration of the first dose of study drug must be planned to take place within 48 hours of moderate or severe ARDS diagnosis
4. Patient is intubated and mechanically ventilated
5. A signed informed consent form from the patient or the patient's personal legal representative or a professional legal representative must be available
6. Patient is aged ≥18 years

Exclusion Criteria:

1. Woman known to be pregnant, lactating or with a positive (urine or serum test) or indeterminate (serum test) pregnancy test
2. Patient is simultaneously taking part in another pharmacotherapy protocol
3. Patient is not expected to survive for 24 hours
4. Patient has an underlying clinical condition where, in the opinion of the Investigator, it would be extremely unlikely that the patient would come off ventilation, e.g., motor neurone disease, Duchenne muscular dystrophy or rapidly progressive interstitial pulmonary fibrosis
5. Patient has severe chronic obstructive pulmonary disease requiring long-term home oxygen therapy or mechanical ventilation (non-invasive ventilation or via tracheotomy) except for continuous positive airway pressure (CPAP) or bi-level positive airway pressure used solely for sleep-disordered breathing
6. Patient has congestive heart failure, defined as New York Heart Association class IV
7. Patient has acute left ventricular failure
8. Patient has liver failure (Child-Pugh grade C)
9. Patient has received any prior interferon
10. Patient has known hypersensitivity to natural or recombinant IFN beta or to any of the excipients
11. Patient is receiving renal dialysis therapy for chronic renal failure
12. Patient is receiving extra-corporeal membrane oxygenation, high-frequency oscillatory ventilation or any form of extra-corporeal lung support
13. Patient has had any form of mechanical ventilation (invasive or non-invasive, excluding CPAP alone) for longer than 48 hours prior to the diagnosis of ARDS. Non-invasive ventilation has to be continuously applied for at least 12 hours per day in these 48 hours
14. Patient has burns to ≥15% of their total body surface area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Bellingan, MD, Study Director — University College London Hospitals, NHS, London, UK; V Marco Ranieri, Prof. MD, Study Director — Universita La Sapeinza Policlinico Umberto I, Rome, Italy
Locations (71):
- Belgium (6):
  - Erasmus Hospital, Brussels
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - CHU Charleroi Site Hôpital Civil Marie Curie, Lodelinsart
  - CHU Dinant Godinne UCL Namur, Yvoir
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Hospital Usti nad Labem, Ústí nad Labem
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- France (15):
  - Nouvel Hôpital Civil, Strasbourg, Alsace
  - Centre Hospitalier Régional d'Orléans, Orléans, Loiret
  - CHU D'Angers, Angers, Pays de la Loire Region
  - CHU De Poitiers, Poitiers, Poitou-Charentes
  - Hôpital de la Croix Rousse, Lyon, Rhône
  - Hôpital Charles-Nicolle, Rouen, Seine-Maritime
  - CHU Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Le Mans, Le Mans
  - Hôpital Nord AP-HM, Marseille
  - CHRU Nancy, Nancy
  - Pitié-Salpêtrière Hospital, Paris
  - CHU Pontchaillou, Rennes
  - CHU Bretonneau, Tours
  - Hôpital Cochin, Réanimation Médicale Hospitalisation, Paris, Île-de-France Region
- Germany (8):
  - Klinikum Augsburg Klinik für Anästhesiologie, Augsburg
  - Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn Klinik und Poliklinik für Anästhesiologie, Bonn
  - Kliniken der Stadt Köln Klinikum Merheim, Cologne
  - Universitätsklinikum Carl Gustav Carus Klinik für Anästhesiologie und Intensivmedizin, Dresden
  - Universitätsmedizin Göttingen Klinik für Anästhesiologie, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Intesivmedizin, Hamburg
  - Universitätsklinik Leipzig Klinik und Poliklinik für Anäesthesiologie und Intensivtherapie, Leipzig
- Italy (6):
  - Azienda Ospedaliera Universitaria Sant' Anna, Cona
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Monza, Monza
  - Universita degli Studi di Roma "La Sapienza", Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - AOU Città della Salute e della Scienza di Torino, Torino
- Spain (15):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario del Henares, Coslada
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario de Gran Canaria Dr Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Corporació Sanitària Parc Taulí, Sabadell
  - Hospital Universitari Mútua de Terrassa, Terrassa
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
- United Kingdom (14):
  - Bristol Royal Infirmary University Hospitals, Bristol Foundation Trust, Bristol
  - University Hospital of Wales, Cardiff
  - Royal Infirmary of Edinburgh, Edinburgh
  - University College London Hospitals, NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St George's University Hospitals, NHS Foundation Trust, London
  - Hammersmith Hospital Imperial College Healthcre NHS Trust, London
  - Charing Cross Hospital St Mary's Hospital, Imperial College Healthcare NHS Trust, London
  - Charing Cross Hospital Imperial College Healthcare NHS Trust, London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Lancashire Treaching Hospitals NHS Foundation Trust, Preston
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jalkanen J, Khan S, Elima K, Huttunen T, Wang N, Hollmen M, Elo LL, Jalkanen S. Polymorphism in interferon alpha/beta receptor contributes to glucocorticoid response and outcome of ARDS and COVID-19. Crit Care. 2023 Mar 16;27(1):112. doi: 10.1186/s13054-023-04388-8. PMID 36927455
- [Derived] Ranieri VM, Pettila V, Karvonen MK, Jalkanen J, Nightingale P, Brealey D, Mancebo J, Ferrer R, Mercat A, Patroniti N, Quintel M, Vincent JL, Okkonen M, Meziani F, Bellani G, MacCallum N, Creteur J, Kluge S, Artigas-Raventos A, Maksimow M, Piippo I, Elima K, Jalkanen S, Jalkanen M, Bellingan G; INTEREST Study Group. Effect of Intravenous Interferon beta-1a on Death and Days Free From Mechanical Ventilation Among Patients With Moderate to Severe Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2020 Feb 25;323(8):725-733. doi: 10.1001/jama.2019.22525. PMID 32065831

RESULTS

PARTICIPANT FLOW:
Groups:
- FP-1201-lyo 10 μg: FP-1201-lyo 10 μg (Interferon beta-1a) will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational product is lyophilisate for solution for injection which will be reconstituted in water for injection.
  Interferon beta-1a: Investigational drug
- Placebo: Placebo will be administered once daily as an intravenous bolus injection for 6 days.
  Investigational placebo product is lyophilisate for solution for injection which will be reconstituted in water for injection.
  Placebo: Placebo for investigational drug
Period: Overall Study
Arm/Group | FP-1201-lyo 10 μg | Placebo
Started (Subjects that received atleast 1 dose of study treatment) | 144 | 152
Subjects Randomised | 146 | 155
Short-Term Follow-Up (Day 28) | 105 | 115
Long-Term Follow-Up (Day 90) | 96 | 101
Long-Term Follow-Up (Day 180) (The study was terminated early) | 73 | 74
Completed (Extended Follow-Up (Day 360), but study was terminated early) | 51 | 49
Not Completed | 93 | 103
Not completed — Death | 51 | 53
Not completed — Lost to Follow-UP, withdrawal of consent | 4 | 7
Not completed — Early termination of study | 38 | 43

BASELINE CHARACTERISTICS:
Population: A total of 296 subjects received at least 1 dose of study treatment (301 subjects fulfilled all criteria and were randomly assigned in a 1:1 ratio to FP-1201-lyo and placebo, but 5 subjects were not dosed).The Full Analysis Set (FAS) consisted of the 296 randomised and treated subjects who received 1 or more doses study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | FP-1201-lyo 10 μg | Placebo | Total
Number analyzed (Participants) | 144 | 152 | 296
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 101 | 190
  >=65 years | 55 | 51 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (17.2) | 58.4 (14.0) | 58.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 61 | 103
  Male | 102 | 91 | 193
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaskan | 1 | 1 | 2
  Race: Native Arab | 4 | 2 | 6
  Race: Asian-Other | 1 | 2 | 3
  Race: Black | 4 | 5 | 9
  Race: Other or not reported | 35 | 36 | 71
  Race: White | 99 | 106 | 205
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 12 | 12 | 24
  Czechia | 1 | 1 | 2
  Finland | 15 | 15 | 30
  Italy | 18 | 19 | 37
  United Kingdom | 25 | 29 | 54
  France | 54 | 58 | 112
  Germany | 8 | 7 | 15
  Spain | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint (VFDsurv; All-cause Mortality and Number of Days Free of Mechanical Ventilation) at Day 28
Description: VFDsurv is a composite measure of all-cause mortality and the number of days free of mechanical ventilation (VFDsurv) within 28 days among survivors. Ventilator-free days (VFDs) correspond to those days when unassisted breathing (UAB) was possible for a complete calendar day. UAB was defined as: spontaneously breathing with face mask, nasal prong oxygen or room air, T-piece breathing, tracheostomy mask breathing, CPAP less than or equal to 5 cmH2O without pressure support or intermittent mandatory ventilation assistance, use of CPAP or BIPAP solely for sleep apnoea management. A patient was reported as ventilator-free after 2 consecutive calendar days of unassisted breathing (a VFD value of 0 is assigned to patients who die without initiating UAB or who require more than 28 days of mechanical ventilation. All patients who die before Day28 are assigned a VFDsurv value of -1).
Time Frame: Day 28
Population: Full Analysis Set (FAS), 296 subjects.
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 10 [-1 to 26] | 8.5 [-1 to 26]
Statistical Analysis 1: Comparison: FP-1201-lyo 10 μg vs Placebo; A non-parametric analysis has been used as the data distribution was skewed. This involved a generalised Wilcoxon rank sum-based stratification test which assigns ranks within strata and compares two treatments within strata (Van Elteren hypothesis test); Test type: Superiority; p = 0.8219, Van Elteren hypothesis test

2. Secondary Outcome: Efficacy Endpoint: All-cause Mortality
Description: Fatalities, mortality all-causes from randomisation up to Day 28
Time Frame: At Day 28
Population: Full Analysis Set (FAS) defined as all randomised subjects that received atleast one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- FP-1201-lyo 10 μg: FP-1201-lyo 10 μg (Interferon beta-1a) for 6 days.
- Placebo: Placebo for 6 days.
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
percentage of subjects | 26.4 [19 to 34] | 23 [17 to 31]

3. Secondary Outcome: Efficacy Endpoint: Mortality in ICU
Description: All-cause mortality for subjects who died in Intensive Care Units up to Day 28.
Time Frame: Up to Day 28
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
percentage of subjects | 25.7 [19 to 34] | 23.0 [17 to 31]

4. Secondary Outcome: Efficacy Endpoint: Mortality in Hospital
Description: This is the number of subjects who died in hospital (i.e. outside of Intensive Care Units) up to Day 28.
Time Frame: Up to Day 28
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Participants | 1 | 0

5. Secondary Outcome: Other Secondary Efficacy Endpoints: Days Free of Organ Failure
Description: The total number of days free of organ failure by Sequential Organ Failure Assessment (SOFA) methodology. Overall, the median number of days free of organ failure was 0 days in both the treatment groups.
Time Frame: Day 28 or last day in intensive care unit [ICU] if patient has left the ICU earlier than Day 28
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 0 [0 to 28] | 0 [0 to 28]

6. Secondary Outcome: Other Secondary Efficacy Endpoints: Days Free of Renal Support
Description: Days without renal support (any renal support was documented). Overall, the median number of days free of renal support was 28 days in the active group and 27 days in the placebo group.
Time Frame: Day 28
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 28 [0 to 28] | 27 [0 to 28]

7. Secondary Outcome: Other Secondary Efficacy Endpoints: Days Free of Vasoactive Support
Description: Days without vasoactive support. The vasoactive support included catecholamine and non-catecholamine vasopressors, inotropes and vasodilating agents.
  Overall, the median number of days free of vasoactive support was 20 days in the active group and 21 days in the placebo group.
Time Frame: Day 28
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 20 [0 to 28] | 21 [1 to 28]

8. Secondary Outcome: Other Secondary Efficacy Endpoint: Days Free of Mechanical Ventilation
Description: The total number of days free of mechanical ventilation has been derived from the Patient Status report recorded on each day during the 28-day period. Patients who died during this period have been assigned a value of zero. This variable differs from the calculated "Ventilation Free Days (VFD) endpoint, which contribute to the VDFsurv primary efficacy endpoint as it require additional conditions of unassisted breathing (UAB) to be met.
Time Frame: Day 28
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 10 [0 to 26] | 9 [0 to 26]
Statistical Analysis 1: Comparison: FP-1201-lyo 10 μg vs Placebo; Van Elteren hypothesis test was used as the distribution was non-normal and negatively skewed by patients who are assigned scores of zero in the event of death; Test type: Superiority; p = 0.4678, Van Elteren p-values

9. Secondary Outcome: Other Secondary Efficacy Endpoints: Number of ICU-free Days
Description: Number of Intensive Care Unit free days up to Day 28, i.e. the patient is no longer receiving care in ICU. Patients who die during this period have been assigned a value of zero for the number of ICU care free days.
Time Frame: Day 28
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 6 [0 to 24] | 3.5 [0 to 24]

10. Secondary Outcome: Other Secondary Efficacy Endpoints: Number of Days in Hospital
Description: Hospitalisation days (including the stay at Intensive Care Units). Patients who died during this period have been assigned a value of 28 for the number of days in ICU or in hospital.
Time Frame: Day 28
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Days | 28 [8 to 28] | 28 [8 to 28]

11. Secondary Outcome: Evaluation of Safety: Adverse Events and Deaths
Description: Adverse events (AE) up to Day 28. Per protocol, AEs occurring after Day 28 if the investigator considered a causal relationship with the study drug as well as all deaths up to Day 360 were reported. Treatment-emergent AEs (TEAEs) were defined as AEs that begins or worsens in intensity after at least one dose of study drug has been administered. Serious AEs (SAEs) were defined as any untoward medical occurrence that at any dose resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was an important medical event.
Time Frame: AEs up to Day 28, only related after Day 28 and deaths up to Day 360
Population: The analysis population included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Participants
  Subjects with TEAE | 130 | 132
  Subjects with AE considered related to study drug | 41 | 33
  Subjects with SAE | 77 | 77
  Death | 51 | 53

12. Secondary Outcome: Efficacy Endpoint: Presence of Neutralising Antibodies to IFN Beta-1a
Description: The immunological response to FP-1201-lyo was assessed by monitoring presence of anti-drug binding antibodies (BAbs) and neutralising antibodies (NAbs) to IFN beta-1a on pre-dose Day 1 and at Day 28, the last day in ICU or early termination (if earlier). The BAbs were determined first, and if present, the NAbs were also determined. Presence of BAbs and NAbs were summarised categorically, using positive/negative classification.
Time Frame: Baseline and Day 28 (or last day in intensive care unit [ICU] or at withdrawal, if earlier)
Population: Full Analysis Set, the subjects who had laboratory evaluation done. Subjects were analysed for IFN beta NAbs only if BAbs were present.
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 142 | 148
Participants
  Presence of BAbs to IFN β-1a at baseline | 2 | 2
  Presence of BAbs to IFN β-1a at Day28 | 0 | 1
  Presence of NAbs to IFN β-1a at baseline | 1 | 0
  Presence of NAbs to IFN β-1a at Day28 | 0 | 0

13. Secondary Outcome: Efficacy Endpoint: Evaluation of Pharmacodynamic (PD) Using Myxovirus Resistance Protein A (MxA) Biomarker
Description: Evaluation of MxA biomarker change from baseline to D14 between treatments arms over time.
Time Frame: From baseline to Day 14
Population: Subjects from Full Analysis Set population for whom samples were available; analysis of last observation performed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 137 | 143
ng/ml | 31.8 (63.3) | 7.8 (28.8)
Statistical Analysis 1: Comparison: FP-1201-lyo 10 μg; Test type: Superiority; p < 0.05, ANCOVA; Analysis of covariance (ANCOVA) model using Type III sums of squares with Treatment, Severity, and Country fixed effect factors, Baseline as covariate

14. Secondary Outcome: Long-term Efficacy Endpoint: Change in Quality of Life From Baseline to Day 180
Description: Quality of Life was assessed through EQ-5D-3L (EuroQol 5-Dimensions 3-Levels questionnaire). An EQ Visual Analogue Scale (VAS) total score (ranging from 0-100) was measured (0= Worst imaginable health state, 100= Best imaginable health state). The EQ-5D-3L VAS scores are numerically summarised as change from pre-dose (Day 1) to long term follow-up (Day 180 visit).
Time Frame: Change from baseline to Day 180
Population: Subjects from Full Analysis Set population who completed QoL questionnaire at Baseline and Day 180.
Measure: Median (Full Range); unit: change score on a scale
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 53 | 43
change score on a scale | -10 [-55 to 70] | -5 [-60 to 91]

15. Secondary Outcome: Long-term Efficacy Endpoints Relating to Respiratory Functioning (FEV1)
Description: Measuring FEV1 (forced expiratory volume in 1 second) assessed pulmonary function (airway obstruction, bronchoconstriction or bronchodilation). FEV1 is the volume exhaled during the first second of a forced expiratory manoeuvre, starting from the level of total lung capacity.
Time Frame: Day 180
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: %FEV1
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 48 | 45
%FEV1 | 81.2 (21.1) | 79.5 (29.6)

16. Secondary Outcome: Long-term Efficacy Endpoints Relating to Neurological Functioning (6MWT)
Description: The 6-minute walk test (6MWT) measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. According to the ERS/ATS technical standard to which the 6MWT was done, the walk test is done twice and the best result is used. It is an evaluation of the global and integrated responses of all systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood and neuromuscular units and muscle metabolism. The self-paced 6MWT assesses the sub- maximal level of functional capacity and will better reflect the functional exercise level for daily activities. ANOVA parameters estimates (LS Means and 90 % conf.interval) for the overall treatment difference was analysed.
Time Frame: Day 180
Population: All subjects in Full Analysis Set population who performed atleast one 6MWT test at Day 180 visit. Furthest distance walked during the two tests was analysed using an ANOVA model.
Measure: Mean (Standard Deviation); unit: maximum distance walked (meters)
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 48 | 45
maximum distance walked (meters) | 449 (174) | 424 (156)
Statistical Analysis 1: Comparison: FP-1201-lyo 10 μg vs Placebo; Treatment effect was analysed using ANOVA parameter estimates (Least Squares Means and 95% Confidence Intervals) for the overall treatment difference for maximum distance walked on Day 180; Test type: Other; p > 0.05, ANOVA; Least Squares Mean = 31.1, 95% CI 2-sided [-37.7 to 99.9]

17. Other Pre Specified Outcome: Evaluation of Safety: Vital Signs - Heart Rate
Description: Vital signs were measured supine pre-dose on Day 1 (baseline) and daily up to Day 28 while the patient was in the ICU. The results at baseline and at last observation performed (LOP) were summarized overall by treatment, variable and time point.
  No statistical analyses were made for vital signs.
Time Frame: From baseline to Last Observation Performed (Day 28 or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Safety Population - no statistical analyses were made for vital signs.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
bpm
  Heart Rate, bpm : Pre-Dose | 93.4 (22.2) | 94.8 (22.5)
  Heart Rate, bpm : LOP | 92.5 (18.3) | 92.7 (19.0)

18. Other Pre Specified Outcome: Evaluation of Safety: Vital Signs - Body Temperature
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Safety Population - no statistical analyses were made for vital signs.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
degrees Celsius
  Body Temperature, degrees C : Pre-Dose | 37.1 (1.1) | 37.2 (1.1)
  Body Temperature, degrees C : LOP | 36.9 (0.9) | 36.8 (0.7)

19. Other Pre Specified Outcome: Evaluation of Safety: Vital Signs - Blood Pressure
Description: as for outcome 17
Time Frame: as for outcome 17
Population: Safety Population - no statistical analyses were made for vital signs.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
mmHg
  Systolic Blood Pressure, mmHg: Pre-Dose | 114.6 (20.4) | 110.2 (18.0)
  Systolic Blood Pressure, mmHg : LOP | 124.3 (22.8) | 120.3 (26.2)
  Diastolic Blood Pressure, mmHg : Pre-Dose | 58.9 (12.9) | 55.6 (9.7)
  Diastolic Blood Pressure, mmHg : LOP | 65.1 (14.8) | 62.6 (13.8)
  Mean Arterial Pressure, mmHg : Pre-Dose | 76.5 (13.9) | 73.6 (11.2)
  Mean Arterial Pressure, mmHg : LOP | 82.7 (15.5) | 80.8 (16.6)

20. Other Pre Specified Outcome: Evaluation of Safety: Physical Examination
Description: Physical examination data (covering the major body systems; general appearance, head [ear, nose and throat], cardiovascular, eyes, respiratory, abdomen, urogenital, musculoskeletal, neurological, lymph nodes and skin) were categorized as "normal"; "abnormal, not clinically significant;" "abnormal, clinically significant" or "not done". Physical examinations were performed at Screening, then at the Last day in ICU and Day 28 (Out of ICU) or Early Termination, from which the last observation performed is derived. The changes from baseline to the last observations performed are categorized as "no change", "change clinically significant"; "change not clinically significant", "not done".
Time Frame: From baseline to Last Observation Performed (D28 or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Safety population - no statistical analyses were made
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Participants
  General Appearance: No change | 59 | 66
  General Appearance: Change, Clinically Significant | 8 | 9
  General Appearance: Change, Not Clinically Significant | 8 | 8
  General Appearance: Not done | 33 | 34
  General Appearance: Not available/pt died | 36 | 35
  Ear, Nose and Throat: No change | 67 | 75
  Ear, Nose and Throat: Change, Clinically Significant | 2 | 1
  Ear, Nose and Throat: Change, Not Clinically Significant | 5 | 6
  Ear, Nose and Throat: Not done | 34 | 35
  Ear, Nose and Throat: Not available/pt died | 36 | 35
  Eyes: No change | 70 | 76
  Eyes: Change, Clinically Significant | 1 | 1
  Eyes: Change, Not Clinically Significant | 2 | 3
  Eyes: Not done | 35 | 36
  Eyes: Not available/pt died | 36 | 36
  Respiratory: No change | 27 | 30
  Respiratory: Change, Clinically Significant | 30 | 28
  Respiratory: Change, Not Clinically Significant | 21 | 26
  Respiratory: Not done | 30 | 33
  Respiratory: Not available/pt died | 36 | 35
  Abdomen: No change | 65 | 70
  Abdomen: Change, Clinically Significant | 3 | 2
  Abdomen: Change, Not Clinically Significant | 9 | 10
  Abdomen: Not done | 31 | 35
  Abdomen: Not available/pt died | 36 | 35
  Urogenital: No change | 67 | 72
  Urogenital: Change, Clinically Significant | 3 | 3
  Urogenital: Change, Not Clinically Significant | 6 | 4
  Urogenital: Not done | 32 | 38
  Urogenital: Not available/pt died | 36 | 35
  Musculoskeletal: No change | 59 | 63
  Musculoskeletal: Change, Clinically Significant | 11 | 8
  Musculoskeletal: Change, Not Clinically Significant | 5 | 9
  Musculoskeletal: Not done | 33 | 37
  Musculoskeletal: Not available/pt died | 36 | 35
  Neurological: No change | 49 | 55
  Neurological: Change, Clinically Significant | 18 | 14
  Neurological: Change, Not Clinically Significant | 8 | 13
  Neurological: Not done | 33 | 34
  Neurological: Not available/pt died | 36 | 36
  Lymph nodes: No change | 69 | 78
  Lymph nodes: Change, Clinically Significant | 0 | 0
  Lymph nodes: Change, Not Clinically Significant | 0 | 0
  Lymph nodes: Not done | 39 | 39
  Lymph nodes: Not available/pt died | 36 | 35
  Skin: No change | 64 | 64
  Skin: Change, Clinically Significant | 3 | 8
  Skin: Change, Not Clinically Significant | 5 | 8
  Skin: Not done | 36 | 37
  Skin: Not available/pt died | 36 | 35
  Cardiovascular: No change | 56 | 60
  Cardiovascular: Change, Clinically Significant | 9 | 8
  Cardiovascular: Change, Not Clinically Significant | 8 | 12
  Cardiovascular: Not done | 33 | 37
  Cardiovascular: Not available/pt died | 38 | 35

21. Other Pre Specified Outcome: Evaluation of Safety: Laboratory Results
Description: Laboratory safety assessments of biochemistry, haematology and urinalysis were performed daily during the stay at ICU. Laboratory data were classified according to normal ranges as out of range (OOR; not clinically significant), OOR (clinically significant), or OOR (clinically significant and an AE). Laboratory test results were summarised by actual results by baseline and last observation period.
Time Frame: From baseline to Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Safety Population -no statistical analyses were made
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Participants
  Haemoglobin, Pre-Dose: Normal | 22 | 30
  Haemoglobin, Pre-Dose: OOR (NCS) | 103 | 107
  Haemoglobin, Pre-Dose: OOR (CS) | 19 | 14
  Haemoglobin, Pre-Dose: OOR (CS+AE) | 0 | 0
  Haemoglobin, Pre-Dose: Not available/pt died | 0 | 1
  Haemoglobin, LOP: Normal | 17 | 18
  Haemoglobin, LOP: OOR (NCS) | 100 | 117
  Haemoglobin, LOP: OOR (CS) | 23 | 16
  Haemoglobin, LOP: OOR (CS+AE) | 3 | 1
  Haemoglobin, LOP: Not available/pt died | 1 | 0
  Platelets, Pre-Dose: Normal | 85 | 91
  Platelets, Pre-Dose: OOR (NCS) | 43 | 42
  Platelets, Pre-Dose: OOR (CS) | 16 | 17
  Platelets, Pre-Dose: OOR (CS+AE) | 0 | 0
  Platelets, Pre-Dose: Not available/pt died | 0 | 2
  Platelets, LOP: Normal | 76 | 65
  Platelets, LOP: OOR (NCS) | 52 | 72
  Platelets, LOP: OOR (CS) | 10 | 10
  Platelets, LOP: OOR (CS+AE) | 5 | 5
  Platelets, LOP: Not available/pt died | 1 | 0
  Leucocytes, Pre-Dose: Normal | 40 | 58
  Leucocytes, Pre-Dose: OOR (NCS) | 72 | 56
  Leucocytes, Pre-Dose: OOR (CS) | 32 | 36
  Leucocytes, Pre-Dose: OOR (CS+AE) | 0 | 0
  Leucocytes, Pre-Dose: Not available/pt died | 0 | 2
  Leucocytes, LOP: Normal | 72 | 57
  Leucocytes, LOP: OOR (NCS) | 52 | 70
  Leucocytes, LOP: OOR (CS) | 15 | 21
  Leucocytes, LOP: OOR (CS+AE) | 3 | 4
  Leucocytes, LOP: Not available/pt died | 2 | 0
  Albumin, Pre-Dose: Normal | 17 | 17
  Albumin, Pre-Dose: OOR (NCS) | 83 | 106
  Albumin, Pre-Dose: OOR (CS) | 20 | 14
  Albumin, Pre-Dose: OOR (CS+AE) | 0 | 0
  Albumin, Pre-Dose: Not available/pt died | 24 | 15
  Albumin, LOP: Normal | 26 | 25
  Albumin, LOP: OOR (NCS) | 97 | 117
  Albumin, LOP: OOR (CS) | 18 | 9
  Albumin, LOP: OOR (CS+AE) | 1 | 0
  Albumin, LOP: Not available/pt died | 2 | 1
  Creatine Kinase, Pre-Dose: Normal | 59 | 62
  Creatine Kinase, Pre-Dose: OOR (NCS) | 32 | 45
  Creatine Kinase, Pre-Dose: OOR (CS) | 19 | 11
  Creatine Kinase, Pre-Dose: OOR (CS+AE) | 1 | 0
  Creatine Kinase, Pre-Dose: Not available/pt died | 33 | 34
  Creatine Kinase, LOP: Normal | 82 | 93
  Creatine Kinase, LOP: OOR (NCS) | 45 | 45
  Creatine Kinase, LOP: OOR (CS) | 11 | 8
  Creatine Kinase, LOP: OOR (CS+AE) | 2 | 0
  Creatine Kinase, LOP: Not available/pt died | 4 | 6
  Creatinine, Pre-Dose: Normal | 78 | 72
  Creatinine, Pre-Dose: OOR (NCS) | 41 | 50
  Creatinine, Pre-Dose: OOR (CS) | 23 | 28
  Creatinine, Pre-Dose: OOR (CS+AE) | 2 | 0
  Creatinine, Pre-Dose: Not available/pt died | 0 | 2
  Creatinine, LOP: Normal | 69 | 73
  Creatinine, LOP: OOR (NCS) | 56 | 64
  Creatinine, LOP: OOR (CS) | 13 | 14
  Creatinine, LOP: OOR (CS+AE) | 5 | 1
  Creatinine, LOP: Not available/pt died | 1 | 0
  Glucose, Pre-Dose: Normal | 56 | 53
  Glucose, Pre-Dose: OOR (NCS) | 76 | 85
  Glucose, Pre-Dose: OOR (CS) | 11 | 10
  Glucose, Pre-Dose: OOR (CS+AE) | 0 | 0
  Glucose, Pre-Dose: Not available/pt died | 1 | 4
  Glucose, LOP: Normal | 65 | 74
  Glucose, LOP: OOR (NCS) | 71 | 75
  Glucose, LOP: OOR (CS) | 7 | 3
  Glucose, LOP: OOR (CS+AE) | 0 | 0
  Glucose, LOP: Not available/pt died | 1 | 0
  Bilirubin, Pre-Dose: Normal | 88 | 106
  Bilirubin, Pre-Dose: OOR (NCS) | 37 | 33
  Bilirubin, Pre-Dose: OOR (CS) | 9 | 6
  Bilirubin, Pre-Dose: OOR (CS+AE) | 0 | 0
  Bilirubin, Pre-Dose: Not available/pt died | 10 | 7
  Bilirubin, LOP: Normal | 114 | 121
  Bilirubin, LOP: OOR (NCS) | 19 | 23
  Bilirubin, LOP: OOR (CS) | 4 | 3
  Bilirubin, LOP: OOR (CS+AE) | 6 | 5
  Bilirubin, LOP: Not available/pt died | 1 | 0
  AST, Pre-Dose: Normal | 57 | 52
  AST, Pre-Dose: OOR (NCS) | 50 | 70
  AST, Pre-Dose: OOR (CS) | 18 | 14
  AST, Pre-Dose: OOR (CS+AE) | 2 | 0
  AST, Pre-Dose: Not available/pt died | 17 | 16
  AST, LOP: Normal | 67 | 76
  AST, LOP: OOR (NCS) | 54 | 56
  AST, LOP: OOR (CS) | 8 | 11
  AST, LOP: OOR (CS+AE) | 11 | 7
  AST, LOP: Not available/pt died | 4 | 2
  ALT, Pre-Dose: Normal | 86 | 92
  ALT, Pre-Dose: OOR (NCS) | 37 | 43
  ALT, Pre-Dose: OOR (CS) | 9 | 9
  ALT, Pre-Dose: OOR (CS+AE) | 2 | 0
  ALT, Pre-Dose: Not available/pt died | 10 | 8
  ALT, LOP: Normal | 72 | 85
  ALT, LOP: OOR (NCS) | 52 | 46
  ALT, LOP: OOR (CS) | 8 | 12
  ALT, LOP: OOR (CS+AE) | 10 | 8
  ALT, LOP: Not available/pt died | 2 | 1
  Bicarbonate, Pre-Dose: Normal | 90 | 97
  Bicarbonate, Pre-Dose: OOR (NCS) | 44 | 47
  Bicarbonate, Pre-Dose: OOR (CS) | 8 | 7
  Bicarbonate, Pre-Dose: OOR (CS+AE) | 0 | 0
  Bicarbonate, Pre-Dose: Not available/pt died | 2 | 1
  Bicarbonate, LOP: Normal | 89 | 105
  Bicarbonate, LOP: OOR (NCS) | 47 | 41
  Bicarbonate, LOP: OOR (CS) | 7 | 6
  Bicarbonate, LOP: OOR (CS+AE) | 0 | 0
  Bicarbonate, LOP: Not available/pt died | 1 | 0
  Urine Protein, Pre-Dose: Normal | 52 | 54
  Urine Protein, Pre-Dose: OOR (NCS) | 67 | 73
  Urine Protein, Pre-Dose: OOR (CS) | 5 | 7
  Urine Protein, Pre-Dose: OOR (CS+AE) | 0 | 0
  Urine Protein, Pre-Dose: Not available/pt died | 20 | 18
  Urine Protein, LOP: Normal | 66 | 84
  Urine Protein, LOP: OOR (NCS) | 63 | 53
  Urine Protein, LOP: OOR (CS) | 10 | 7
  Urine Protein, LOP: OOR (CS+AE) | 0 | 1
  Urine Protein, LOP: Not available/pt died | 5 | 7
  Urine Glucose, Pre-Dose: Normal | 114 | 123
  Urine Glucose, Pre-Dose: OOR (NCS) | 9 | 7
  Urine Glucose, Pre-Dose: OOR (CS) | 0 | 3
  Urine Glucose, Pre-Dose: OOR (CS+AE) | 0 | 0
  Urine Glucose, Pre-Dose: Not available/pt died | 21 | 19
  Urine Glucose, LOP: Normal | 128 | 135
  Urine Glucose, LOP: OOR (NCS) | 9 | 10
  Urine Glucose, LOP: OOR (CS) | 1 | 0
  Urine Glucose, LOP: OOR (CS+AE) | 0 | 0
  Urine Glucose, LOP: Not available/pt died | 6 | 7
  Urine Blood, Pre-Dose: Normal | 48 | 53
  Urine Blood, Pre-Dose: OOR (NCS) | 67 | 75
  Urine Blood, Pre-Dose: OOR (CS) | 10 | 8
  Urine Blood, Pre-Dose: OOR (CS+AE) | 0 | 0
  Urine Blood, Pre-Dose: Not available/pt died | 19 | 16
  Urine Blood, LOP: Normal | 57 | 58
  Urine Blood, LOP: OOR (NCS) | 73 | 77
  Urine Blood, LOP: OOR (CS) | 9 | 10
  Urine Blood, LOP: OOR (CS+AE) | 0 | 0
  Urine Blood, LOP: Not available/pt died | 5 | 7

22. Other Pre Specified Outcome: Evaluation of Pharmacoeconomics: Days Free of Organ Failure
Description: Due to the study terminating early, costs items from hospitals were not collected and pharmacoeconomic analyses could not be done.
Time Frame: Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Costs items from hospitals were not collected.
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 0 | 0

23. Other Pre Specified Outcome: Evaluation of Pharmacoeconomics: Days Free of Renal Support
Description: as for outcome 22
Time Frame: Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Costs items from hospitals were not collected.
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 0 | 0

24. Other Pre Specified Outcome: Evaluation of Pharmacoeconomics: Days Free of Vasoactive Support
Description: as for outcome 22
Time Frame: Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Costs items from hospitals were not collected.
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 0 | 0

25. Other Pre Specified Outcome: Evaluation of Pharmacoeconomics: Days Free of Mechanical Ventilation
Description: as for outcome 22
Time Frame: Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Costs items from hospitals were not collected
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: Evaluation of Pharmacoeconomics: Number of ICU-free Days
Description: as for outcome 22
Time Frame: Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Costs items from hospitals were not collected
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 0 | 0

27. Other Pre Specified Outcome: Evaluation of Pharmacoeconomics: Number of Days in Hospital
Description: as for outcome 22
Time Frame: Day 28 (or last day in ICU if patient has left the ICU earlier than Day 28, or at withdrawal)
Population: Costs items from hospitals were not collected.
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 0 | 0

28. Other Pre Specified Outcome: Exploratory Variables Relating to Efficacy: Composite Endpoint (Mortality and Days Free of Mechanical Ventilation) at Day 90
Description: Composite endpoint including mortality and days free of mechanical ventilation (VFDsurv) within 90 days among survivors. Ventilation Free Survival at Day 90 has been classified as Dead, Alive but on a ventilator and Alive and breathing unassisted
Time Frame: Within 90 days
Population: Full Analysis Set (discontinued not included).
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Participants
  Dead | 47 | 48
  Alive-on ventilator | 6 | 10
  Alive-breathing unassisted | 90 | 91

29. Other Pre Specified Outcome: Change in the Treatment-specific Exploratory Biomarker Cluster of Differentiation 73 (CD73) Concentration
Description: Evaluation of Cluster of differentiation 73 (CD73) change from baseline to D14 between treatments arms over time.
Time Frame: From baseline to Day 14
Population: Subjects from Full Analysis Set population for whom samples were available; analysis of last observation performed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 141 | 148
ng/ml | 6.2 (8.9) | 6.1 (7.9)

30. Other Pre Specified Outcome: Changes in Levels of Potential Inflammatory Markers (PIMs)
Description: Evaluation of potential inflammatory markers (PIMs) change from baseline to D14 between treatments arms over time. Potential biomarkers included IL-1ra, IL-6, FGF basic, IP-10 and TNF-α.
Time Frame: From baseline to Day 14
Population: Subjects from Full Analysis Set population for whom samples were available; analysis of last observation performed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 142 | 149
pg/mL
  IL-1ra | 1830 (5252) | 1699 (4565)
  IL-6 | 63 (298) | 88 (584)
  FGF basic | 37 (17) | 38 (20)
  IP-10 | 1938 (3543) | 1762 (3894)
  TNF-α | 68 (60) | 81 (148)
Statistical Analysis 1: Comparison: FP-1201-lyo 10 μg; IL -1ra - changes in levels from baseline to Day 14; Test type: Other; p > 0.05, ANCOVA; ANCOVA estimates (LS means and a 95 % CI for the treatment difference) were presented for all numeric biomarker variables; LS Means difference = 0
Statistical Analysis 2: Comparison: FP-1201-lyo 10 μg; IL- 6 - changes in levels from baseline to Day 14; Test type: Other; p > 0.05, ANCOVA; [statistical method as in outcome 30, analysis 1]; LS Means difference = 0
Statistical Analysis 3: Comparison: FP-1201-lyo 10 μg; FGF basic - changes in levels from baseline to Day 14; Test type: Other; p < 0.05, ANCOVA; ANCOVA estimates (LS means and a 95% CI for the treatment difference) were presented for all numeric biomarker variables; LS Means difference = 0
Statistical Analysis 4: Comparison: FP-1201-lyo 10 μg; IP-10 - changes in levels from baseline to Day 14; Test type: Other; p < 0.05, ANCOVA; [statistical method as in outcome 30, analysis 1]; LS Means difference = 0
Statistical Analysis 5: Comparison: FP-1201-lyo 10 μg; TNF-α - changes in levels from baseline to Day 14; Test type: Other; p > 0.05, ANCOVA; [statistical method as in outcome 30, analysis 1]; LS Means difference = 0

31. Other Pre Specified Outcome: Pharmacogenetic Analysis
Description: An optional genetic sample was analysed for subjects based on a separate consent. A carrier frequency was analysed for a C/T polymorphism (rs9984723) located in the 3'PRIME_UTR/intron region of IFNAR2-gene, which encodes the beta chain for the IFN-alpha/beta receptor and encompasses a regulatory motif for the glucocorticoid receptor. Biomarker responders were defined by a 3-fold elevation in MxA and a 2-fold in CD73 in comparison to baseline.
Time Frame: Anytime from baseline to Day 28
Population: Only subjects with consent for a genetic sample were analysed. Carriers of the C-allele were analysed in biomarker responders compared to biomarker non-responders. 5 and 6 subjects failed to provide genotype information in analyses for responder and non-responders, respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Biomarker Responder; Biomarker Non-responder: FP-1201-lyo 10 μg (Interferon beta-1a) for 6 days.
Arm/Group | Biomarker Responder | Biomarker Non-responder
Number analyzed (Participants) | 38 | 79
Participants
  C-allele carrier | 21 | 26
  C-allele non-carrier | 12 | 47
Statistical Analysis 1: Comparison: Biomarker Responder; Test type: Other; p < 0.007, Chi-squared — The p-value is not adjusted for multiple comparisons

32. Other Pre Specified Outcome: Exploratory, Extended Long-term Follow-up: Overall Mortality at Day 360
Description: Fatalities; as the study was terminated early, the assessment time point for mortality at Day 360 was not reached. Therefore only the overall mortality at study termination is presented.
Time Frame: Day 360 /termination of study
Population: Full Analysis Set, but the study was terminated early. The mortality numbers include 3 study subjects who had SAEs with an onset before the first dose of IMP and who subsequently died.
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
Participants | 51 | 53

33. Other Pre Specified Outcome: Extended Long-term Follow-up Exploratory Endpoint: Change in Quality of Life From Baseline to Day 360
Description: Quality of Life was assessed through EQ-5D-3L (EuroQol 5-Dimensions 3-Levels questionnaire). An EQ Visual Analogue Scale (VAS) total score (ranging from 0-100) was measured (0= Worst imaginable health state, 100= Best imaginable health state). The EQ-5D-3L VAS scores are numerically summarised as change from pre-dose (Day 1) to extended long term follow-up (Day 360 visit).
Time Frame: Change from baseline to Day 360
Population: Subjects from Full Analysis Set population who completed QoL questionnaire at Baseline and Day 360. As the study was terminated early, only a limited amount of data were available at the post-baseline time point.
Measure: Median (Full Range); unit: change score on a scale
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 37 | 33
change score on a scale | 0 [-59 to 35] | 0 [-80 to 86]

34. Other Pre Specified Outcome: Neurological Functioning (6MWT) at Extended Long-term Follow-up
Description: The 6-minute walk test (6MWT) measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. According to the ERS/ATS technical standard to which the 6MWT was done, the walk test is done twice and the best result is used. It is an evaluation of the global and integrated responses of all systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood and neuromuscular units and muscle metabolism. The self-paced 6MWT assesses the sub- maximal level of functional capacity and will better reflect the functional exercise level for daily activities. ANOVA parameters estimates (LS Means and 90 % confidence intervals) for the overall treatment difference was analysed.
Time Frame: Day 360
Population: All subjects in Full Analysis Set population who performed atleast one 6MWT test at Day 360, before the study was early terminated.
Measure: Mean (Standard Deviation); unit: maximal distance walked (meters)
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 32 | 31
maximal distance walked (meters) | 475 (119) | 453 (190)
Statistical Analysis 1: Comparison: FP-1201-lyo 10 μg vs Placebo; Treatment effect was analysed using ANOVA parameter estimates (Least Squares Means and 95 % Confidence Intervals) for the overall treatment difference for maximun distance walked on Day 360; Test type: Other; p > 0.05, ANOVA; Least Squares Mean = 28, 95% CI 2-sided [-54 to 110.1]

35. Other Pre Specified Outcome: Extended Long-term Follow-up Endpoint: Respiratory Functioning (FEV1) at Day 360
Description: as for outcome 15
Time Frame: Day 360
Population: Subjects from Full Analysis Set population attending Day 360 visit.
Measure: Mean (Standard Deviation); unit: %FEV1
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 33 | 27
%FEV1 | 69.4 (31.8) | 72.0 (28.5)

36. Post Hoc Outcome: Post-Hoc Analyses Related to the Use of Concomitant Glucocorticoids Medications and Mortality at D28
Description: The overall use of concomitant glucocorticoids treatment in both study treatment groups (active and placebo) were analysed.
Time Frame: Day 28
Population: Subjects who received at least 1 dose of concomitant glucocorticoids during days 0-28
Measure: Number; unit: percentage of participants
Arm/Group | FP-1201-lyo 10 μg | Placebo
Number analyzed (Participants) | 144 | 152
percentage of participants
  Use of concomitant glucocorticoids: number analyzed (Participants) | 78 | 98
  Use of concomitant glucocorticoids | 54.1 | 64.5
  Mortality, with concomitant glucocorticoids: number analyzed (Participants) | 78 | 98
  Mortality, with concomitant glucocorticoids | 39.7 | 27.6
  Mortality, without concomitant glucocorticoids: number analyzed (Participants) | 66 | 54
  Mortality, without concomitant glucocorticoids | 10.6 | 14.8

ADVERSE EVENTS:
Time Frame: The Adverse Event (AE) reporting period extended up to study Day 28. In accordance with the protocol, the investigators reported AEs occurring after Day 28 only if the investigator considered a causal relationship with the study drug. All deaths were reported as SAEs throughout the study, up until Day 360.
Description: The "Serious Adverse Event" list and the "Other (Not including Serious) Adverse Event" list present all reported Treatment Emergent Adverse Events (defined as an AE that begins or that worsens in severity after at least one dose of study drug). In 3 study subjects a non-treatment emergent SAE began before first dose of the study drug (included in mortality numbers because these SAEs led to death )
Arm/Group | FP-1201-lyo 10 μg | Placebo
All-Cause Mortality (participants affected / at risk) | 51/144 | 53/152
Serious Adverse Events (participants affected / at risk) | 77/144 | 77/152
Other Adverse Events (participants affected / at risk) | 109/144 | 110/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-1201-lyo 10 μg (N=144) | Placebo (N=152)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 13 (13) | 8 (8)
CONDITION AGGRAVATED (General disorders) | 7 (7) | 11 (12)
DISEASE PROGRESSION (General disorders) | 3 (3) | 1 (1)
DEATH (General disorders) | 1 (1) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
BRAIN DEATH (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 9 (9)
SEPTIC SHOCK (Infections and infestations) | 7 (7) | 5 (5)
SEPSIS (Infections and infestations) | 2 (2) | 4 (4)
BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1)
EMPYEMA (Infections and infestations) | 2 (2) | 0 (0)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER MENINGOENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
MENINGITIS ASPERGILLUS (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SYSTEMIC CANDIDA (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 6 (6) | 2 (2)
SHOCK (Vascular disorders) | 2 (2) | 4 (4)
HYPERTENSION (Vascular disorders) | 4 (4) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 4 (4) | 5 (5)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 2 (2)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC DISORDER (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 (1) | 0 (0)
TORSADE DE POINTES (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 3 (3) | 2 (2)
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
BRAIN HYPOXIA (Nervous system disorders) | 1 (1) | 0 (0)
BRAIN INJURY (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL VENOUS THROMBOSIS (Nervous system disorders) | 0 (0) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
QUADRIPLEGIA (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 (2) | 2 (2)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADENOCARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DIFFUSE LARGE B-CELL LYMPHOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO KIDNEY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROENDOCRINE CARCINOMA OF THE SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 5 (5)
POST INFECTION GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 0 (0)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BAROTRAUMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DELAYED RECOVERY FROM ANAESTHESIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GASTROINTESTINAL ANASTOMOTIC COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RENAL REPLACEMENT THERAPY (Surgical and medical procedures) | 0 (0) | 2 (2)
WITHDRAWAL OF LIFE SUPPORT (Surgical and medical procedures) | 1 (1) | 1 (1)
EXTRACORPOREAL MEMBRANE OXYGENATION (Surgical and medical procedures) | 0 (0) | 1 (1)
GASTRIC OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
LAPAROTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 2 (2) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BIOPSY BONE MARROW ABNORMAL (Investigations) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2) | 0 (0)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1)
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-1201-lyo 10 μg (N=144) | Placebo (N=152)
PNEUMONIA (Infections and infestations) | 8 (8) | 4 (4)
SEPTIC SHOCK (Infections and infestations) | 1 (2) | 3 (4)
SEPSIS (Infections and infestations) | 8 (8) | 3 (3)
BACTERAEMIA (Infections and infestations) | 3 (3) | 5 (5)
DEVICE RELATED SEPSIS (Infections and infestations) | 3 (3) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1) | 2 (2)
FUNGAL INFECTION (Infections and infestations) | 2 (2) | 1 (1)
INFECTION (Infections and infestations) | 2 (2) | 1 (1)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (2) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 2 (2) | 0 (0)
ENTEROBACTER PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2)
IMPETIGO (Infections and infestations) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 (1) | 0 (0)
SUPERINFECTION (Infections and infestations) | 1 (1) | 1 (1)
SYSTEMIC CANDIDA (Infections and infestations) | 0 (0) | 1 (1)
ASPERGILLUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL DISEASE CARRIER (Infections and infestations) | 1 (1) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 1 (1)
CANDIDA PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
CANDIDURIA (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
EPIGLOTTITIS (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
FUNGAEMIA (Infections and infestations) | 1 (1) | 0 (0)
GENITAL HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1)
HERPES SIMPLEX PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
LYMPHANGITIS (Infections and infestations) | 1 (1) | 0 (0)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0)
OTITIS MEDIA ACUTE (Infections and infestations) | 1 (1) | 0 (0)
PANCREATIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
RENAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SPUTUM PURULENT (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
THROMBOPHLEBITIS SEPTIC (Infections and infestations) | 1 (1) | 0 (0)
TINEA CRURIS (Infections and infestations) | 1 (1) | 0 (0)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
VULVOVAGINITIS (Infections and infestations) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (8)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
INCREASED BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LARYNGEAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY ALKALOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 17 (21) | 12 (12)
CONDITION AGGRAVATED (General disorders) | 3 (3) | 5 (5)
CHILLS (General disorders) | 2 (4) | 0 (0)
GENERALISED OEDEMA (General disorders) | 2 (2) | 3 (3)
HYPERTHERMIA (General disorders) | 1 (1) | 2 (2)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 (2) | 1 (1)
HYPOTHERMIA (General disorders) | 0 (0) | 2 (2)
MEDICAL DEVICE COMPLICATION (General disorders) | 1 (1) | 1 (1)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 1 (1)
CATHETER SITE NECROSIS (General disorders) | 1 (1) | 0 (0)
DISEASE RECURRENCE (General disorders) | 0 (0) | 1 (1)
DRUG WITHDRAWAL SYNDROME (General disorders) | 1 (1) | 0 (0)
HYPERTHERMIA MALIGNANT (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 11 (12) | 14 (14)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 7 (7)
VOMITING (Gastrointestinal disorders) | 4 (4) | 5 (5)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 2 (2) | 4 (4)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 2 (2) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 2 (2)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 1 (1)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 2 (2)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
ABDOMINAL COMPARTMENT SYNDROME (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
REGURGITATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 9 (11) | 15 (16)
TACHYCARDIA (Cardiac disorders) | 2 (2) | 6 (6)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 (4) | 3 (3)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 3 (3)
CARDIAC DISORDER (Cardiac disorders) | 1 (1) | 1 (1)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 (2) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CYANOSIS (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 9 (10) | 7 (7)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 8 (9) | 4 (5)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (5) | 6 (9)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
ALKALOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
MALNUTRITION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERAMMONAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OVERWEIGHT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 11 (13) | 10 (10)
SHOCK HAEMORRHAGIC (Vascular disorders) | 2 (2) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1) | 6 (6)
VENOUS THROMBOSIS (Vascular disorders) | 4 (4) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 1 (1)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 1 (1) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1)
PHLEBITIS (Vascular disorders) | 0 (0) | 1 (1)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 (0) | 1 (1)
VASCULAR OCCLUSION (Vascular disorders) | 0 (0) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 2 (2) | 7 (9)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 5 (5)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2) | 4 (4)
HEPATIC ENZYME INCREASED (Investigations) | 2 (2) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CHLORIDE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD LACTIC ACID INCREASED (Investigations) | 0 (0) | 2 (2)
BLOOD POTASSIUM INCREASED (Investigations) | 2 (2) | 0 (0)
BLOOD SODIUM INCREASED (Investigations) | 1 (1) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 2 (2)
ANTICOAGULATION DRUG LEVEL INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD GLUCOSE DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD IRON DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1)
CLOSTRIDIUM TEST POSITIVE (Investigations) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 (1) | 0 (0)
ELECTROENCEPHALOGRAM ABNORMAL (Investigations) | 0 (0) | 1 (1)
EOSINOPHIL COUNT INCREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
MYOGLOBIN BLOOD INCREASED (Investigations) | 1 (1) | 0 (0)
PO2 DECREASED (Investigations) | 0 (0) | 1 (1)
RED BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
SPLEEN SCAN ABNORMAL (Investigations) | 1 (1) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 16 (18) | 11 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 7 (7) | 6 (6)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
COAGULOPATHY (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HISTIOCYTOSIS HAEMATOPHAGIC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 9 (9) | 8 (8)
CHOLESTASIS (Hepatobiliary disorders) | 3 (3) | 5 (5)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 4 (4) | 3 (3)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 3 (3) | 3 (3)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 2 (2)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 6 (7) | 7 (7)
DELIRIUM (Psychiatric disorders) | 8 (8) | 3 (3)
ANXIETY (Psychiatric disorders) | 4 (4) | 2 (2)
INSOMNIA (Psychiatric disorders) | 3 (3) | 2 (2)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0)
WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 (1) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 1 (1) | 0 (0)
NIGHTMARE (Psychiatric disorders) | 0 (0) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 7 (8) | 8 (8)
RENAL FAILURE (Renal and urinary disorders) | 6 (6) | 5 (5)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 1 (2)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 2 (2)
RENAL INJURY (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 3 (3) | 7 (7)
CONFUSIONAL STATE (Nervous system disorders) | 1 (1) | 2 (2)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 2 (2) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SEDATION (Nervous system disorders) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
ENDOTRACHEAL INTUBATION COMPLICATION (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
BAROTRAUMA (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
TRACHEAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
EAR INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOREIGN BODY ASPIRATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MECHANICAL VENTILATION COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MIXED CONNECTIVE TISSUE DISEASE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RENAL REPLACEMENT THERAPY (Surgical and medical procedures) | 1 (1) | 2 (2)
ENDOTRACHEAL INTUBATION (Surgical and medical procedures) | 0 (0) | 2 (2)
EXTRACORPOREAL MEMBRANE OXYGENATION (Surgical and medical procedures) | 0 (0) | 1 (1)
GASTRECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTROSTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
TRACHEOSTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CONJUNCTIVAL OEDEMA (Eye disorders) | 2 (2) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 1 (1) | 0 (0)
EYE DISORDER (Eye disorders) | 0 (0) | 1 (1)
PUPILS UNEQUAL (Eye disorders) | 1 (1) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 1 (1)
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
As the study was terminated early, only a limited amount of data was available at Day 180 and Day 360.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT02622724/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02622724/SAP_001.pdf